CLINICAL TRIAL: NCT04183192
Title: Pharmacodynamic Biomarkers to Support Biosimilar Development: Clinical Study 1: Interleukin-5 Antagonists - Mepolizumab and Reslizumab
Brief Title: Pharmacodynamic Biomarkers to Support Biosimilar Development: Interleukin-5 Antagonists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SCR-006
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Healthy Subjects; Pharmacokinetics; Pharmacodynamics
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — mepolizumab; reslizumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of four dose groups (low, intermediate low, intermediate high, and high) of each drug (mepolizumab or reslizumab) or placebo
Who Masked: Participant, Investigator
Masking Description: The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing.
  Subjects and staff will be blinded to treatment assignment during confinement, but route of administration will not be blinded. The blind will be maintained through a randomization schedule held by the dispensing pharmacist. Subjects and staff will be informed of a subject's end of study day when discharged from confinement. Subjects and staff will not be informed of the specific treatment arm assignment. The clinical research nurse will administer the study drugs in unit dose containers that are not transparent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Arm A: Mepolizumab low dose (Experimental): Single dose of mepolizumab 3 mg SC
  Interventions: Biological: Mepolizumab
- Arm B: Mepolizumab low intermediate dose (Experimental): Single dose of mepolizumab 6 mg SC
  Interventions: Biological: Mepolizumab
- Arm C: Mepolizumab high intermediate dose (Experimental): Single dose of mepolizumab 12 mg SC
  Interventions: Biological: Mepolizumab
- Arm D: Mepolizumab high dose (Experimental): Single dose of mepolizumab 24 mg SC
  Interventions: Biological: Mepolizumab
- Arm E: Reslizumab low dose (Experimental): Single dose of reslizumab 0.1 mg/kg IV
  Interventions: Biological: Reslizumab
- Arm F: Reslizumab intermediate low dose (Experimental): Single dose of reslizumab 0.2 mg/kg IV
  Interventions: Biological: Reslizumab
- Arm G: Reslizumab high intermediate dose (Experimental): Single dose of reslizumab 0.4 mg/kg IV
  Interventions: Biological: Reslizumab
- Arm H: Reslizumab high dose (Experimental): Single dose of reslizumab 0.8 mg/kg IV
  Interventions: Biological: Reslizumab
- Arm I: Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab 3 mg administered SC
  Arms: Arm A: Mepolizumab low dose
Biological: Mepolizumab — Mepolizumab 6 mg administered SC
  Arms: Arm B: Mepolizumab low intermediate dose
Biological: Mepolizumab — Mepolizumab 12 mg administered SC
  Arms: Arm C: Mepolizumab high intermediate dose
Biological: Mepolizumab — Mepolizumab 24 mg administered SC
  Arms: Arm D: Mepolizumab high dose
Biological: Reslizumab — Reslizumab 0.1 mg/kg administered IV
  Arms: Arm E: Reslizumab low dose
Biological: Reslizumab — Reslizumab 0.2 mg/kg administered IV
  Arms: Arm F: Reslizumab intermediate low dose
Biological: Reslizumab — Reslizumab 0.4 mg/kg administered IV
  Arms: Arm G: Reslizumab high intermediate dose
Biological: Reslizumab — Reslizumab 0.8 mg/kg administered IV
  Arms: Arm H: Reslizumab high dose
Biological: Placebo — Placebo (administered either IV or SC)
  Arms: Arm I: Placebo

SUMMARY:
This study is designed to assess pharmacokinetics and pharmacodynamics of mepolizumab and reslizumab across an appropriate dose range to inform clinical trial operating characteristics for future clinical pharmacology pharmacodynamics similarity studies.

This is a randomized, placebo-controlled, single-dose, parallel arm study in 72 healthy subjects assigned to one of four dose groups (low, intermediate low, intermediate high, and high) of each drug (mepolizumab or reslizumab) or placebo.

DETAILED DESCRIPTION:
This study is designed to assess pharmacokinetics and pharmacodynamics of mepolizumab and reslizumab across an appropriate dose range to inform clinical trial operating characteristics for future clinical pharmacology pharmacodynamics similarity studies.

This is a randomized, placebo-controlled, single-dose, parallel arm study in 72 healthy subjects assigned to one of four dose groups (low, intermediate low, intermediate high, and high) of each drug (mepolizumab or reslizumab) or placebo. Mepolizumab doses are 3, 6, 12, or 24 mg. Reslizumab doses are 0.1, 0.2, 0.4, or 0.8 mg/kg. Each arm will include 8 subjects (4 male and 4 female).

Subjects will be admitted for treatment on day -1 and receive a single dose of study drug or placebo on day 1. Depending on the treatment arm, subjects will remain in confinement for two weeks and continue follow-up through either day 63 or day 123.

Blood samples (approximately 5 mL per sample) will be collected for determination of plasma concentrations for study drug. Additional blood samples will be collected for determination of eosinophil counts (5 mL per sample; pharmacodynamic measure) and exploratory proteomics analyses (5 mL per sample).

Safety evaluations will include adverse event (AE) monitoring, vital sign measurements, and physical examinations. All AEs reported by the subject or observed by the investigator or clinical research unit (CRU) staff will be recorded. Any AE reported after the informed consent is signed and before study drug application will be recorded as medical history.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an institutional review board approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 55 years of age, inclusive, who has a body mass index of 18.5 to 29.9 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and Check-in (Day -1).
5. Subject has a peripheral blood eosinophil count of ≥50 and ≤700 cells per microliter of blood as measured by a standard hematology analyzer.
6. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before Check in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day -1) until at least 1 month after the end of the study.
7. Male subjects must agree to practice 1 highly effective method of birth control (as determined by the investigator or designee) from at least 1 month before Check in (Day -1) until at least 1 month after the end of the study.
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study

Exclusion Criteria:

1. Subject is taking any medication known to affect leukocyte population numbers.
2. Subject is anemic (i.e., with Hct or Hgb less than the lower limit of normal) or has any chronic condition(s) that may impact blood sample collection.
3. Subject has had previous exposure to the biologic mepolizumab or reslizumab.
4. Subject has a history of asthma.
5. Subject has a history of anaphylaxis from environmental exposures such as peanuts or bee stings.
6. Subject has an allergic history that includes urticaria, angioedema or respiratory coughing or bronchospasm.
7. Subject has a history of severe local reactions or generalized erythema from skin allergen testing.
8. Subject is anemic or has any chronic condition(s) that may impact blood sample collection.
9. Subject has used any prescription or nonprescription drugs (including aspirin or NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug.
10. Subjects are currently participating in another clinical study of an investigational drug or are have been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
11. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks of Screening.
12. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, chocolate, cola), caffeine, grapefruit, or grapefruit juice within 48 hours of dosing. Subjects must refrain from ingesting these throughout the study.
13. Subject has any underlying disease or surgical or medical condition (e.g., cancer, human immunodeficiency virus [HIV], severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study. This includes subjects with any underlying medical conditions that put subjects at higher risk for coronavirus disease of 2019 (COVID-19) complications; per current Center for Disease Control and Prevention (CDC) recommendations this includes:

    * People with chronic lung disease or moderate to severe asthma
    * People who have serious heart conditions
    * People who are immunocompromised
    * Many conditions can cause a person to be immunocompromised, including cancer treatment, smoking, bone marrow or organ transplantation, immune deficiencies, poorly controlled HIV, and prolonged use of corticosteroids and other immune weakening medications
    * People with severe obesity (body mass index [BMI] of 40 or higher)
    * People with diabetes
    * People with chronic kidney disease undergoing dialysis
    * People with liver disease
14. Subject has any signs or symptoms that are consistent with COVID-19. Per current CDC recommendations this includes subjects with the symptoms cough or shortness of breath or difficulty breathing, or at least two of the following symptoms: fever, chills, repeated shaking with chills, muscle pain, headache, sore throat or new loss of taste/smell. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
15. Subject tests positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by a molecular diagnostic test performed prior to admission.
16. Subject has known or suspected allergies or sensitivities to any study drug.
17. Subject has clinical laboratory test results (hematology, serum chemistry) at Screening that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
18. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
19. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
20. Female subjects are pregnant or lactating before enrollment in the study.
21. Subject is known to have, or is suspected to have, a parasitic infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Deering, MSN, APNP, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as a part of manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as any eventual publications.
Supporting Information: Study Protocol, SAP
Time Frame: April, 2022. Materials will be available indefinitely.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Mepolizumab Low Dose | Arm B: Mepolizumab Low Intermediate Dose | Arm C: Mepolizumab High Intermediate Dose | Arm D: Mepolizumab High Dose | Arm E: Reslizumab Low Dose | Arm F: Reslizumab Intermediate Low Dose | Arm G: Reslizumab High Intermediate Dose | Arm H: Reslizumab High Dose | Arm I: Placebo
Started | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Mepolizumab Low Dose | Arm B: Mepolizumab Low Intermediate Dose | Arm C: Mepolizumab High Intermediate Dose | Arm D: Mepolizumab High Dose | Arm E: Reslizumab Low Dose | Arm F: Reslizumab Intermediate Low Dose | Arm G: Reslizumab High Intermediate Dose | Arm H: Reslizumab High Dose | Arm I: Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [25 to 50] | 29 [23 to 45] | 33 [28 to 50] | 39 [34 to 42] | 46 [35 to 52] | 36 [31 to 41] | 45 [28 to 50] | 49 [33 to 51] | 40 [30 to 52] | 39 [28 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 3 | 2 | 2 | 2 | 2 | 2 | 21
  Male | 5 | 6 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 9
  Not Hispanic or Latino | 6 | 8 | 7 | 7 | 8 | 6 | 7 | 7 | 7 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 6 | 4 | 5 | 3 | 3 | 2 | 3 | 33
  White | 3 | 5 | 2 | 4 | 3 | 2 | 3 | 6 | 5 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 72
Body Weight [Median (Inter-Quartile Range); unit: kg] | 73 [68 to 81] | 71 [67 to 82] | 72 [68 to 81] | 79 [66 to 84] | 75 [67 to 85] | 80 [75 to 84] | 78 [73 to 87] | 72 [67 to 80] | 82 [73 to 84] | 77 [68 to 84]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 25.3 [23.6 to 27.8] | 23.7 [22.9 to 27.4] | 26.7 [24.6 to 28.4] | 24.8 [24.0 to 26.3] | 23.9 [22.4 to 26.6] | 27.5 [24.2 to 28.9] | 26.2 [24.5 to 28.2] | 23.8 [22.1 to 26.9] | 27.5 [24.4 to 29.1] | 25.6 [23.0 to 28.1]

OUTCOME MEASURES:

1. Primary Outcome: Area Under Effect Curve (AUEC) for Eosinophils for Mepolizumab and Reslizumab
Description: The values and variability of AUEC for eosinophils at low, intermediate low, intermediate high, and high doses of mepolizumab and reslizumab. AUEC was calculated as percentage change from baseline and used all measures from time zero to the last sample collected on study. Calculations were performed using non-compartmental analysis packages available in R software.
Time Frame: Day -1 and 0h (pre-dose), 24h (post-dose); once daily from Day 2 onwards until Day 14 post-dose; once weekly from Day 21 onwards until Day 63 post-dose for Arms A, B, E, F and until Day 123 post-dose for Arms C, D, G, H, and I.
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline * day
Arm/Group | Arm A: Mepolizumab Low Dose | Arm B: Mepolizumab Low Intermediate Dose | Arm C: Mepolizumab High Intermediate Dose | Arm D: Mepolizumab High Dose | Arm E: Reslizumab Low Dose | Arm F: Reslizumab Intermediate Low Dose | Arm G: Reslizumab High Intermediate Dose | Arm H: Reslizumab High Dose | Arm I: Placebo
Number analyzed (Participants) | 7 | 8 | 7 | 7 | 8 | 8 | 8 | 8 | 8
Percentage change from baseline * day | -1804 (1425) | -195 (1568) | -1456 (1951) | -1428 (2442) | -1748 (1888) | -1075 (1312) | -3313 (4506) | -2905 (1423) | -1409 (3410)

2. Primary Outcome: Maximum Change From Baseline for Eosinophils for Mepolizumab and Reslizumab
Description: The values and variability of maximal change from baseline for eosinophils at low, intermediate low, intermediate high, and high doses of mepolizumab and reslizumab. Values are percentage change from baseline.
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Arm A: Mepolizumab Low Dose | Arm B: Mepolizumab Low Intermediate Dose | Arm C: Mepolizumab High Intermediate Dose | Arm D: Mepolizumab High Dose | Arm E: Reslizumab Low Dose | Arm F: Reslizumab Intermediate Low Dose | Arm G: Reslizumab High Intermediate Dose | Arm H: Reslizumab High Dose | Arm I: Placebo
Number analyzed (Participants) | 7 | 8 | 7 | 7 | 8 | 8 | 8 | 8 | 8
Percentage change from baseline | -72 (73) | -63 (14) | -82 (23) | -85 (14) | -79 (9) | -67 (27) | -75 (25) | -77 (25) | -41 (15)

3. Secondary Outcome: Maximum Concentration (Cmax) for Mepolizumab and Reslizumab
Description: The values and variability of Cmax at low, intermediate low, intermediate high, and high doses of mepolizumab and reslizumab.
Time Frame: 0 (pre-dose), 1, 4, 12, 24, hours post-dose; once daily from Day 3 onwards until Day 14 post-dose; once weekly from Day 21 onwards until Day 63 post-dose for Arms A, B, E, F and until Day 123 post-dose for Arms C, D, G, and H.
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm A: Mepolizumab Low Dose | Arm B: Mepolizumab Low Intermediate Dose | Arm C: Mepolizumab High Intermediate Dose | Arm D: Mepolizumab High Dose | Arm E: Reslizumab Low Dose | Arm F: Reslizumab Intermediate Low Dose | Arm G: Reslizumab High Intermediate Dose | Arm H: Reslizumab High Dose
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 5 | 8 | 8 | 8
μg/mL | 0.36 (74) | 0.53 (54) | 1.21 (23) | 2.05 (27) | 3.1 (10) | 5.2 (35) | 12.3 (26) | 18.7 (20)

4. Secondary Outcome: Area Under the Curve (AUC) for Mepolizumab and Reslizumab
Description: The values and variability of AUC at low, intermediate low, intermediate high, and high doses of mepolizumab and reslizumab.
Time Frame: as for outcome 3
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL*day
Arm/Group | Arm A: Mepolizumab Low Dose | Arm B: Mepolizumab Low Intermediate Dose | Arm C: Mepolizumab High Intermediate Dose | Arm D: Mepolizumab High Dose | Arm E: Reslizumab Low Dose | Arm F: Reslizumab Intermediate Low Dose | Arm G: Reslizumab High Intermediate Dose | Arm H: Reslizumab High Dose
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 5 | 8 | 8 | 8
μg/mL*day | 17.6 (73) | 21.7 (153) | 38.1 (21) | 61.8 (46) | 150 (109) | 152 (239) | 450 (72) | 420 (70)

5. Secondary Outcome: Pharmacodynamic Model Parameters (Maximum Effect [Emax]) for Eosinophil Area Under the Effect Curve Versus Dose Emax Models for Mepolizumab or Reslizumab
Description: The model parameter (Emax, units percentage change from baseline * day) from an Emax model for eosinophil area under the effect curve versus dose were calculated after combining data from low, intermediate low, intermediate high, and high doses of mepolizumab or reslizumab with placebo data. AUEC (units of percentage change from baseline * day) was calculated as percentage change from baseline and used all measures from time zero to the last sample collected on study. Model-analyses were conducted using the DoseFinding package available in R software. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 2500 repetitions.
Time Frame: as for outcome 1
Population: Analysis population for each group was limited to those subjects administered mepolizumab or placebo (the mepolizumab group) or administered reslizumab or placebo (reslizumab group) who completed the study. Results from subjects administered placebo were used in all analyses.
Measure: Mean (95% Confidence Interval); unit: Percentage change from baseline * day
Groups:
- Mepolizumab: Area Under the Effect Curve Model for Eosinophils: Model-based analysis using individual subject baseline-subtracted area under the effect curve results from all mepolizumab and placebo arms.
- Reslizumab: Area Under the Effect Curve Model for Eosinophils: Model-based analysis using individual subject baseline-subtracted area under the effect curve results from all reslizumab and placebo arms.
Arm/Group | Mepolizumab: Area Under the Effect Curve Model for Eosinophils | Reslizumab: Area Under the Effect Curve Model for Eosinophils
Number analyzed (Participants) | 38 | 40
Percentage change from baseline * day | 10840 [6571 to 31670] | 10446 [4138 to 22373]

6. Secondary Outcome: Pharmacodynamic Model Parameter, ED50 (Half Maximal Effect Dose), for Eosinophil Area Under the Effect Curve Versus Dose Emax Model for Mepolizumab
Description: The model parameter (ED50, units mg) from an Emax model for eosinophil area under the effect curve versus dose were calculated after combining data from low, intermediate low, intermediate high, and high doses of mepolizumab with placebo data. AUEC (units of percentage change from baseline * day) was calculated as percentage change from baseline and used all measures from time zero to the last sample collected on study. Model-analyses were conducted using the DoseFinding package available in R software. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 2500 repetitions.
Time Frame: Day -1 and 0h (pre-dose), 24h (post-dose); once daily from Day 2 onwards until Day 14 post-dose; once weekly from Day 21 onwards until Day 63 post-dose for Arms A, B, and until Day 123 post-dose for Arms C, D, and I.
Population: Analysis population for each group was limited to those subjects administered mepolizumab or placebo (the mepolizumab group) who completed the study. Results from subjects administered placebo were used in all analyses.
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Mepolizumab: Area Under the Effect Curve Model for Eosinophils
Number analyzed (Participants) | 38
mg | 31.3 [8.6 to 400]

7. Secondary Outcome: Pharmacodynamic Model Parameter, ED50 (Half Maximal Effect Dose), for Eosinophil Area Under the Effect Curve Versus Dose Emax Model for Reslizumab
Description: The model parameter (ED50, units mg/kg) from an Emax model for eosinophil area under the effect curve versus dose were calculated after combining data from low, intermediate low, intermediate high, and high doses of reslizumab with placebo data. AUEC (units of percentage change from baseline * day) was calculated as percentage change from baseline and used all measures from time zero to the last sample collected on study. Model-analyses were conducted using the DoseFinding package available in R software. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 2500 repetitions.
Time Frame: Day -1 and 0h (pre-dose), 24h (post-dose); once daily from Day 2 onwards until Day 14 post-dose; once weekly from Day 21 onwards until Day 63 post-dose for Arms E, F and until Day 123 post-dose for Arms G, H, and I.
Population: Analysis population for each group was limited to those subjects administered reslizumab or placebo (reslizumab group) who completed the study. Results from subjects administered placebo were used in all analyses.
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Reslizumab: Area Under the Effect Curve Model for Eosinophils
Number analyzed (Participants) | 40
mg/kg | 0.31 [0.01 to 1.20]

8. Secondary Outcome: Pharmacodynamic Model Parameters (Maximum Effect [Emax]) for Eosinophil Maximum Change From Baseline Versus Dose Emax Models With Mepolizumab or Reslizumab
Description: The model parameter (Emax, units percentage change from baseline) from an Emax model for eosinophil maximum change from baseline versus dose was calculated after combining data from low, intermediate low, intermediate high, and high doses of mepolizumab or reslizumab with placebo data. Maximum change from baseline (units of percentage change from baseline) was calculated as percentage change from baseline and considered all measures from time zero to the last sample collected on study. Model-analyses were conducted using the DoseFinding package available in R software. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 2500 repetitions.
Time Frame: as for outcome 1
Population: Analysis population for each group was limited to those subjects administered mepolizumab or placebo (the mepolizumab group) or administered reslizumab or placebo (reslizumab) who completed the study. Results from subjects administered placebo were used in all analyses.
Measure: Mean (95% Confidence Interval); unit: Percentage change from baseline
Groups:
- Mepolizumab: Maximum Change From Baseline Model for Eosinophils: Model-based analysis using individual subject baseline-subtracted maximum change from baseline results from all mepolizumab and placebo arms.
- Reslizumab: Maximum Change From Baseline Model for Eosinophils: Model-based analysis using individual subject baseline-subtracted maximum change from baseline results from all reslizumab and placebo arms.
Arm/Group | Mepolizumab: Maximum Change From Baseline Model for Eosinophils | Reslizumab: Maximum Change From Baseline Model for Eosinophils
Number analyzed (Participants) | 38 | 40
Percentage change from baseline | 85 [78 to 92] | 86 [77 to 95]

9. Secondary Outcome: Pharmacodynamic Model Parameter, ED50 (Half Maximal Effect Dose), for Eosinophil Maximum Change From Baseline Curve Versus Dose Emax Model Mepolizumab
Description: The model parameter (ED50, units mg) from an Emax model for eosinophil maximum change from baseline versus dose was calculated after combining data from low, intermediate low, intermediate high, and high doses of mepolizumab with placebo data. Maximum change from baseline (units of percentage change from baseline) was calculated as percentage change from baseline and considered all measures from time zero to the last sample collected on study. Model-analyses were conducted using the DoseFinding package available in R software. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 2500 repetitions.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Mepolizumab: Maximum Change From Baseline Model for Eosinophils
Number analyzed (Participants) | 38
mg | 3.8 [2.0 to 6.4]

10. Secondary Outcome: Pharmacodynamic Model Parameter, ED50 (Half Maximal Effect Dose), for Eosinophil Maximum Change From Baseline Curve Versus Dose Emax Model Reslizumab
Description: The model parameter (ED50, units mg/kg) from an Emax model for eosinophil maximum change from baseline versus dose was calculated after combining data from low, intermediate low, intermediate high, and high doses of reslizumab with placebo data. Maximum change from baseline (units of percentage change from baseline) was calculated as percentage change from baseline and considered all measures from time zero to the last sample collected on study. Model-analyses were conducted using the DoseFinding package available in R software. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 2500 repetitions.
Time Frame: as for outcome 7
Population: Analysis population for each group was limited to those subjects administered reslizumab or placebo (reslizumab) who completed the study. Results from subjects administered placebo were used in all analyses.
Measure: Mean (95% Confidence Interval); unit: mg/kg
Arm/Group | Reslizumab: Maximum Change From Baseline Model for Eosinophils
Number analyzed (Participants) | 40
mg/kg | 0.04 [0.01 to 0.08]

ADVERSE EVENTS:
Time Frame: 63 days for subjects in treatment groups A,B,E,F and 123 days for subjects in treatment groups C,D,G, H.
Arm/Group | Arm A: Mepolizumab Low Dose | Arm B: Mepolizumab Low Intermediate Dose | Arm C: Mepolizumab High Intermediate Dose | Arm D: Mepolizumab High Dose | Arm E: Reslizumab Low Dose | Arm F: Reslizumab Intermediate Low Dose | Arm G: Reslizumab High Intermediate Dose | Arm H: Reslizumab High Dose | Arm I: Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 3/8 | 1/8 | 3/8 | 2/8 | 4/8 | 6/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Mepolizumab Low Dose (N=8) | Arm B: Mepolizumab Low Intermediate Dose (N=8) | Arm C: Mepolizumab High Intermediate Dose (N=8) | Arm D: Mepolizumab High Dose (N=8) | Arm E: Reslizumab Low Dose (N=8) | Arm F: Reslizumab Intermediate Low Dose (N=8) | Arm G: Reslizumab High Intermediate Dose (N=8) | Arm H: Reslizumab High Dose (N=8) | Arm I: Placebo (N=8)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vessel puncture site paresthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT04183192/Prot_001.pdf
  • Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04183192/SAP_002.pdf
  • Informed Consent Form (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT04183192/ICF_000.pdf